CLINICAL TRIAL: NCT01050621
Title: Phase I - II Clinical Trial of Combination Conventional Cytotoxic Chemotherapy and Intravenous Vitamin C in Patients With Advanced Cancer or Hematologic Malignancy for Whom Cytotoxic Chemotherapy Alone is Only Marginally Effective
Brief Title: Trial of Chemotherapy Plus Intravenous Vitamin C in Patients With Advanced Cancer for Whom Chemotherapy Alone is Only Marginally Effective
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, John Hoffer, Physician, Jewish General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VITC-003
Record Dates: First submitted 2010-01-11; First posted 2010-01-15 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Cancer
Keywords: ascorbic acid; vitamin C; antioxidants; redox therapy; cytotoxic chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: vitamin C (ascorbic acid) — ascorbic acid 1.5 g/kg body weight infused over 90 to 120 minutes two or three times weekly concurrent with standard cytotoxic chemotherapy individually selected for each patient by the treating oncologist on the basis of best current clinical practice

SUMMARY:
Concurrent administration of intravenous vitamin C (ascorbic acid, 1.5 g/kg, infused two or three times weekly) together with certain cytotoxic chemotherapy regimens could prove to be an effective treatment for some patients with advanced malignancies for whom existing chemotherapy is usually ineffective. The primary objectives of this study are to identify a tolerable and safe dose of intravenous vitamin C when administered during cytotoxic chemotherapy while attempting to empirically identify specific vitamin C-chemotherapy regimens for which the clinical response is unusually favorable after a minimum of 2 months of therapy, as determined by CT scan and biomarkers, when appropriate.

DETAILED DESCRIPTION:
Cytotoxic chemotherapy is relatively ineffective for a large proportion of common cancers. Combining redox active molecules with certain chemotherapy regimens could increase their anti-cancer activity or protect host tissues from toxicity with no loss of anti-cancer activity. Research in this area has been advocated by cancer organizations, but previous clinical trials of combination chemotherapy and antioxidant therapy been small, poorly designed, and unsystematic. Appropriate study of this treatment concept requires a systematic, meticulous empirical approach similar to the one used in conventional cytotoxic drug discovery. This is a Phase I-II study designed to identify promising chemotherapy-antioxidant protocols and determine their acceptability and limiting toxicity in patients with relentlessly progressive cancers for which conventional chemotherapy is clinically indicated but is known to be minimally or marginally effective.

The tolerable dose of intravenous ascorbic acid (IVAA) for cancer patients with normal renal function not receiving chemotherapy is 1.5 g/kg per 90 to 120 minute infusion (Hoffer et al, Ann Oncol 2008;19:1969-1974). Side effects are minimal to non-existent. In this dose-escalating study the IVAA will be 0.9 g/kg per infusion for the first chemotherapy cycle, increasing to 1.5 g/kg per infusion in subsequent cycles, for the first 3 participants. If well tolerated as expected, the initial dose will be 1.5 g/kg per infusion for subsequent participants. Infusions will take place 2 or 3 times per week, bracketing the days of chemotherapy. Standard tolerance and adverse effect criteria will be used. Therapy will continue for a minimum of 2 months, and continue further in the event of disease stabilization or response, as determined from CT scan and biomarkers, with evaluations continuing every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* must be a resident of Quebec, Canada
* documented advanced or metastatic cancer or hematologic malignancy in adults over age 18, with measurable disease
* adequate bone marrow, hepatic, renal and cardiac function so as to permit conventional chemotherapy
* no current calcium oxalate nephrolithiasis with the potential to reduce urinary flow
* life expectancy at least 8 weeks.

Exclusion Criteria:

* glucose-6-phosphate dehydrogenase deficiency
* cancers for which existing chemotherapy offers more than a 33% likelihood of a clinically meaningful response
* serum creatinine greater than 175 micromol/L
* serious GI diseases
* infections
* recent major surgery
* dementia
* altered mental status or other condition that would preclude chemotherapy, including poor functional status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IV ascorbic acid (IVAA) in target dose of 1500 mg/kg supplementing cytotoxic chemotherapeutic drugs. Standard adverse effect criteria will be used. | At every clinic visit
Observe for qualitative indicators that IV ascorbic acid mitigates chemotherapy adverse effects | Every treatment cycle

SECONDARY OUTCOMES:
To monitor for disease arrest or response (RECIST criteria) in a population in which arrest or response is unusual or rare | CT assessment every 2 months
Quality of life assessment using FACT B and POMS R | every month
Measure the effect of chemotherapy on pharmacokinetics of intravenous ascorbic acid | Before and 5 days following first chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Leonard John Hoffer, MD PhD, Principal Investigator — Faculty of Medicine, McGill University
Locations (1):
- Clinical Research Unit, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hoffer LJ, Robitaille L, Zakarian R, Melnychuk D, Kavan P, Agulnik J, Cohen V, Small D, Miller WH Jr. High-dose intravenous vitamin C combined with cytotoxic chemotherapy in patients with advanced cancer: a phase I-II clinical trial. PLoS One. 2015 Apr 7;10(4):e0120228. doi: 10.1371/journal.pone.0120228. eCollection 2015. PMID 25848948